CLINICAL TRIAL: NCT00620139
Title: Proximal Molecular Effects of Concurrent Chemoradiotherapy on Head and Neck Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-016
Record Dates: First submitted 2008-01-25; First posted 2008-02-21 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; chemoradiotherapy; molecular effects; 05-016
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Blood Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Some patients presenting with suspicious lesions of the oropharynx or oral cavity will need to undergo transoral biopsy in the clinic to confirm the diagnosis of carcinoma. Of those patients who choose to participate in the study, an extra piece of tumor will be harvested for investigational purposes related to this trial.
  Interventions: Biological: the arachidonic acid and EGFR signaling pathways and their interaction in HNSCC tumorigenesis,

INTERVENTIONS:
Biological: the arachidonic acid and EGFR signaling pathways and their interaction in HNSCC tumorigenesis, — patient will undergo transoral pretreatment biopsy of the tumor. A comparable second tumor biopsy will be performed in the office after exactly 5 days of concurrent CRT (5 daily fractions of 180-200 cGy radiotherapy and a single cycle of Cisplatin or Carboplatin/5-FU based chemotherapy).Blood plasma and single-void urine specimens will be collected contemporaneously,before and after 5 days of concurrent CRT.

SUMMARY:
This pilot study seeks to evaluate the feasibility of measuring the proximal effects of concurrent chemoradiotherapy (CRT) on the expression of potential therapeutic target molecules in Head and Neck Squamous Cell Carcinoma (HNSCC). Specifically, this study proposes to evaluate the extent to which CRT induces the differential expression of components along two critical, and potentially interdependent, molecular pathways: the arachidonic acid and epidermal growth factor receptor (EGFR) signaling pathways.

ELIGIBILITY:
Inclusion Criteria:

* Untreated HNSCC (> Stage I) amenable to transoral biopsy.
* Scheduled for concurrent CRT (Cisplatin or Carboplatin/5-FU based) as definitive primary treatment
* Older than 18 years of age.
* Understand and sign informed consent.

Exclusion Criteria:

* Any prior treatment of the index cancer (chemotherapy, immunotherapy, hormonal therapy or radiation therapy) or similar treatment of an unrelated malignancy within 6 weeks of enrollment into this study.
* Breast-feeding, pregnancy or of childbearing potential (including those women who are less than two years post menopausal) and unable to confirm adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since last menses.
* History of chronic inflammatory disease (e.g. ulcerative colitis, Crohn's disease, rheumatoid arthritis or pancreatitis).
* Corticosteroid use within 6 weeks of enrollment, excluding topical nasal sprays.
* NSAID (including celecoxib) or aspirin (> 81 mg/day) use within 1 week of enrollment.
* Investigational medication use within 6 weeks of enrollment or is scheduled to receive an investigational drug during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the proximal effects of concurrent chemoradiotherapy (CRT) on the expression of potential therapeutic molecular targets along the arachidonic acid and epidermal growth factor receptor (EGFR) signaling pathways in HNSCC. | Conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org